CLINICAL TRIAL: NCT06808269
Title: Prospective Comparative Multicenter Study of the Care Pathway After Shoulder Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Victor Hugo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-28-CVH
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Injury
Keywords: shoulder surgery; pain; comfort
MeSH Terms: conditions — Shoulder Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- structured follow-up after surgery (Experimental)
  Interventions: Procedure: Vivalto Dom follow-up
- liberal follow-up after surgery (Active Comparator)
  Interventions: Procedure: Liberal follow-up

INTERVENTIONS:
Procedure: Vivalto Dom follow-up — During the pre-operative consultation, the patient receives a prescription for medication (analgesics and anti-inflammatories) for immediate post-operative pain relief. They also receive a "patient information booklet" (see appendix 6). On discharge from surgery, the patient returns home with Vivalto Dom in charge of nursing care and follow-up medication.
  Vivalto Dom is a homecare structure whose mission is to coordinate the discharge of patients back home, and to ensure continuity of overall care (care and social aspects) between the hospital and the city.
  Arms: structured follow-up after surgery
Procedure: Liberal follow-up — The pre-operative and operative course (fasting rules, skin preparation, hospitalization, surgery) is the same as for all routine care patients. The patient is informed before surgery that he or she must make an appointment with a nurse for post-operative care at home; a prescription for medication (analgesics and anti-inflammatories) has been given by the anaesthetist for immediate analgesic treatment, and on discharge from hospital he or she receives another prescription from the surgeon for oral relay treatment.
  Follow-up at home takes place over 3 days, with a private nurse visiting the patient's home every day.
  During the follow-up, the nurse performs clinical monitoring of the following items: pulse, blood pressure, temperature, pain, bleeding, monitoring of the surgical wound, transit, nausea and vomiting. The patient is also guided through the medication protocol.
  Arms: liberal follow-up after surgery

SUMMARY:
Post-operative management of shoulder surgery patients, particularly in terms of pain management and follow-up, can vary from one center to another, influencing clinical outcomes and patient satisfaction. The aim of this study is to compare two approaches to post-operative follow-up in two distinct centers: structured follow-up using the Vivalto-Dom protocol in Paris, and autonomous follow-up through contact with a nurse in Saint-Grégoire. The hypothesis is that these differences in the care pathway will affect pain management, comfort and patient satisfaction. By controlling for operative variability (a single surgeon operating in both centers), the study will identify the most effective follow-up practices for improving post-operative management, with the ultimate aim of optimizing quality of care and reducing post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for one of the following 4 types of surgery: Simple non-repair arthroscopic surgery (acromion, calcification), arthroscopic repair surgery (cuff, DAS, bankart), open surgery without prosthesis (ligamentoplasty, bone block), open surgery with prosthesis (inverted prosthesis, anatomic prosthesis, etc.).

Exclusion Criteria:

* Patients with one or more communication disorders.
* Pregnant or breast-feeding patients
* Patients not covered by a social security scheme
* Refusal to participate in research
* Patients unable to understand or give informed consent
* Patients under guardianship, deprived of liberty or under court protection
* Patients with past or present drug addiction
* Patients with neuropathy
* Patients with cognitive disorders
* Patients with chronic illnesses or inflammatory pathologies leading to chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (VAS) | 3 days, 6 weeks, 3 months and 6 months after surgery
  Pain will be measured using VAS (visual analog scale), from 0 ("no pain") to 10 (maximal pain)

SECONDARY OUTCOMES:
Patient comfort (Likert scale) | 3 days, 6 weeks, 3 months and 6 months after surgery
  Patient comfort will be evaluated using a Likert scale for 6 questions. Scale is from 1 (total discomfort) to 5 (total comfort)
Postoperative complications | 3 days, 6 weeks, 3 months and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Victor Hugo, Paris
  - Centre hospitalier privé Saint-Grégoire, Saint-Grégoire

IPD SHARING:
Plan to Share IPD: No